CLINICAL TRIAL: NCT03373565
Title: Snuff-box Deep Palmar Arch Artery Versus Radial Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamidreza Mahboobi (Other)
Responsible Party: Sponsor-Investigator, Hamidreza Mahboobi, Principle Investigator, Hormozgan University of Medical Sciences
Organization: Hormozgan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUMS.REC.1396.82
Record Dates: First submitted 2017-11-18; First posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radial (Active Comparator): Coronary angiography using radial approach
  Interventions: Procedure: Radial
- palmar (Experimental): Coronary angiography using palmar approach
  Interventions: Procedure: Palmar

INTERVENTIONS:
Procedure: Radial — Coronary angiography using radial approach
  Arms: Radial
Procedure: Palmar — Coronary angiography using radial approach
  Arms: palmar

SUMMARY:
Angiography is a common diagnostic and therapeutic procedure in patients with acute coronary syndrome (ACS). The complications are variable between mild self-limited complications to severe life-threatening complications which need early interventions.

New angiographic methods are associated with variable complications. Death, myocardial infarction, and stroke are among major angiography complications. In addition, some local complications including bleeding at the site of insertion, infection, arteriovenous fistula, pseudoaneurysm, and thrombosis is reported after angiography.

Radial and femoral methods are common angiographic methods. Its shown that radial method is associated with less complications and patients need shorter duration of hospitalization.

Radial artery thrombosis is common complication of radial angiography. However, the prevalence is between 5 to 19 percent but often it is not clinically important. Risk of ischemia due to thrombosis is low because of blood flow in radial and ulnar and collaterals. In patients with incomplete palmar arch this is important and may cause ischemia.

The aim of this study is to compare the outcomes of coronary angiography using Snuff-box deep palmar arch artery and radial artery in patients attending angiography center of Shahid Mohammadi hospital in Bandar Abbas in 2017.

ELIGIBILITY:
Inclusion Criteria:

* indication of coronary artery angiography confirmed by a cardiologist
* Accepting to sign the written informed consent

Exclusion Criteria:

* No follow up visit after one-month period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-20 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Thrombosis | 1 months
  Thrombosis at the site of angiography using ultrasonography

SECONDARY OUTCOMES:
Infection | 1 months
  Number of patients with infection at the site of angiography in physical examnination
Pain | 1 months
  Number of patients with pain at the site of angiography using questionnaire
Numbness | 1 months
  Number of patients with numbness at the site of angiography using questionnaire
Loss of movement | 1 months
  Number of patients with loss of movement at the site of angiography in physical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Hormozgan University of Medical Sciences, Bandar Abbas, Hormozgan, Iran

IPD SHARING:
Plan to Share IPD: Undecided